CLINICAL TRIAL: NCT00458211
Title: Evaluation of Efficacy and Tolerability of Switching to Ziprasidone From Other Antipsychotic Medications
Brief Title: Efficacy and Tolerability of Switching to Ziprasidone From Other Antipsychotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bronx Psychiatric Center (Other Government)
Collaborators: Pfizer (Industry); Buffalo Psychiatric Center (Other); Rochester Psychiatric Center (Other)
Responsible Party: Principal Investigator, Nigel Bark MD, Director of Scizophrenia Research, Bronx Psychiatric Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPCIRB 03-02
Record Dates: First submitted 2007-04-06; First posted 2007-04-10 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Ziprasidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Open label change to ziprasidone
  Interventions: Drug: ziprasidone

INTERVENTIONS:
Drug: ziprasidone — Ziprasidone by mouth 40mg twice a day (bid) for one day, then 80mg bid; may be increased to 120mg bid after three weeks

SUMMARY:
Because ziprasidone has not been extensively studied and is not widely accepted in the severely mentally ill in State hospitals this study aims to demonstrate its effectiveness and relative lack of side effects. 75 patients with schizophrenia or schizoaffective disorder who need a change of medication because of ineffectiveness or side effects will be changed to ziprasidone and followed with detailed assessments for eight weeks.

The hypothesis is that they will improve and have fewer side effects.

DETAILED DESCRIPTION:
Ziprasidone has been found in studies and practice to be efficacious and tolerated well but has not been well studied or well accepted in the very severely ill in State Hospitals. This study aims to fill that gap by examining 75 patients with schizophrenia or schizoaffective disorder who require a change of medication because of poor response or unacceptable side effects.

After signing consent and having a baseline assessment they will, if necessary, be reduced to one antipsychotic then started on ziprasidone, increasing to 160mg the second day. The one antipsychotic they had been on will be reduced over a week and stopped. The ziprasidone can be increased to 240mg after three weeks if necessary.

The study will last eight weeks with efficacy assessed by Clinical Global Impressions (CGI), Positive and Negative Syndrome Scale (PANSS) every two weeks and Brief Assessment of Cognition, Calgary Depression Scale for Schizophrenia, Personal Evaluation of Transitions in Treatment and Medical Outcomes Study Cognitive Questions at the beginning and end. Side effects will be measured by movement disorder scales (Simpson-Angus scale for Parkinsonism (SANRS), Abnormal Involuntary Movement Scale (AIMS) and Barnes Akathisia Scale (BAS)), ECG and weight and blood metabolic measures.

The hypothesis is that ziprasidone will be generally effective and that side effects especially metabolic indices will be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or schizoaffective
* Capacity to give consent
* Stable, on the same medication for a month but only partial response or with unacceptable side effects 18-65 years of age

Exclusion Criteria:

* Repeated non-compliance
* Current depot medication
* Active medical conditions
* QTc >500msec
* Previous non-response
* Previous treatment with ziprasidone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Bark, MD, Principal Investigator — Bronx Psychiatric Center; Jeffrey Grace, MD, Principal Investigator — Buffalo Psychiatric Center; Steven Schwarzkopf, MD, Principal Investigator — Rochester Psychiatric Center
Locations (2):
- United States (2):
  - Buffalo Psychiatric Center, Buffalo, New York
  - Bronx Psychiatric Center, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 subjects from three State Hospitals were recruited and participated between 2005 and 2008: four in-patients from Rochester Psychiatric Center, 17 out-patients from Buffalo Psychiatric Center and 19 in-patients from Bronx Psychiatric Center
Groups:
- Experimental: Open label change to ziprasidone up to 120mg twice a day with meals
Period: Overall Study
Arm/Group | Experimental
Started | 40
Completed | 24 (12 early termination 2 protocol violation 2 ( from Rochester) withdrawn from further analysis)
Not Completed | 16
Not completed — Lack of Efficacy | 12
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: The four Rochester subjects were dropped. The 17 Buffalo subjects were all out patients and 20 years older than the 19 Bronx subjects who were all in-patients. Buffalo subjects were 88% white (Bronx 5%), 12% African American (Bronx 39%), 0% Hispanic (Bronx 50%), 24% with Substance abuse (Bronx 68%)
Arm/Group | Experimental
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS) Measuring Symptoms of Schizophrenia
Description: Minimum score 32 (best) maximum 210 (worst)
Time Frame: Baseline to 8 weeks
Population: The four Rochester subjects were dropped as Rochester could not continue the study.19 Bronx and 17 Buffalo subjects were analyzed separately because they were so different(see baseline characteristics)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Experimental
Number analyzed (Participants) | 36
score on scale
  Bronx baseline | 95 (16)
  Bronx end | 99 (25)
  Buffalo baseline | 72 (22)
  Buffalo end | 62 (19)

2. Secondary Outcome: Clinical Global Impression (CGI) Scores the Evaluator's Overall Impression of Severity (CGI-S) or Change (CGI-I) in Illness.
Description: CGI-S scores from 1 = normal to 7 = most extremely ill
Time Frame: 8 weeks
Population: 17 Buffalo subjects and 19 Bronx subjects
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Experimental
Number analyzed (Participants) | 36
score on scale
  Bronx baseline | 4.6 (0.6)
  Bronx end | 4.9 (0.8)
  Buffalo baseline | 3.5 (0.9)
  Buffalo end | 2.8 (0.8)

3. Secondary Outcome: Weight
Time Frame: 8 weeks
Population: Same as PANNS above
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Experimental
Number analyzed (Participants) | 36
pounds
  Bronx baseline | 195 (43)
  Bronx end | 193 (41)
  Buffalo baseline | 213 (57)
  Buffalo end | 204 (52)

4. Secondary Outcome: Fasting Glucose
Description: Amount of glucose in the blood in mg/dl
Time Frame: 8 weeks
Population: See PANSS above
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Experimental
Number analyzed (Participants) | 36
mg/dl
  Bronx baseline | 91 (28)
  Bronx end | 82 (24)
  Buffalo baseline | 94 (18)
  Buffalo end | 93 (19)

5. Secondary Outcome: Cholesterol
Time Frame: 8 weeks
Population: See PANSS above
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental
Number analyzed (Participants) | 36
mg/dL
  Bronx baseline | 185 (44)
  Bronx end | 160 (28)
  Buffalo baseline | 186 (42)
  Buffalo end | 179 (36)

6. Secondary Outcome: Abnormal Involuntary Movement Scale (AIMS) Measures Tardive Dyskinesia
Description: Scores 0 (none) to 4 (severe) choreo-athetoid and dystonic movements of seven parts of the body with a maximum score 28
Time Frame: 8 weeks
Population: 17 Buffalo subjects and 19 Bronx subjects
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Experimental: All subjects, 17 at Buffalo and 19 at Bronx were given Ziprasidone.
Arm/Group | Experimental
Number analyzed (Participants) | 36
score on scale
  Bronx baseline | 0.3 (0.8)
  Bronx end | 0.3 (0.7)
  Buffalo baseline | 2.9 (3.1)
  Buffalo end | 1.6 (1.4)

7. Secondary Outcome: Simpson-Angus Scale Measures Drug Induced Parkinsonism
Description: Measures 10 signs, (not all of which are now considered Parkinsonism), minimum score 0 (no Parkinsonism) maximum 40.
Time Frame: 8 weeks
Population: see PANNS above
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Experimental
Number analyzed (Participants) | 36
score on scale
  Bronx baseline | 0.2 (0.5)
  Bronx end | 0.1 (0.2)
  Buffalo baseline | 3.6 (3.6)
  Buffalo end | 2.5 (2.6)

8. Secondary Outcome: Corrected QT Interval (QTc)
Description: Time interval between Q and T waves on EKG corrected for pulse rate. Over 500 msec may be dangerous
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Experimental
Number analyzed (Participants) | 36
msec
  Bronx baseline | 396 (18)
  Bronx end | 411 (15)
  Buffalo baeline | 412 (21)
  Buffalo end | 427 (17)

9. Secondary Outcome: Brief Assessment of Cognition in Schizophrenia (BACS)
Description: Scores on the BACS scale, which measures cognition, were changed to Z-scores based on normal controls from Keefe (2008) A Z-score of zero would indicate cognition the same as the normal controls. Negative scores indicate cognition worse than the normal. Theoretically there are no maximum or minimum scores.
Time Frame: 8 weeks
Population: The overall number of participants is made up of 17 at Buffalo and 19 in the Bronx
Measure: Mean (Standard Deviation); unit: Z-score from score on scale
Groups:
- Experimental: Open label change to ziprasidone up to 120mg twice a day with meals, 17 at Buffalo, 19 at Bronx
Arm/Group | Experimental
Number analyzed (Participants) | 36
Z-score from score on scale
  Bronx baseline: number analyzed (Participants) | 19
  Bronx baseline | -14 (6.0)
  Bronx end: number analyzed (Participants) | 19
  Bronx end | -13 (5.3)
  Buffalo baseline: number analyzed (Participants) | 17
  Buffalo baseline | -12 (5.9)
  Buffalo end: number analyzed (Participants) | 17
  Buffalo end | -11 (6.5)

10. Secondary Outcome: Calgary Depression Scale for Schizophrenia
Description: Score on scale, from 0 to 27, above 6 considered indicative of depression, higher scores mean worse outcome,
Time Frame: 8 weeks
Population: 19 at Bronx, 17 at Buffalo
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 36
score on a scale
  Bronx baseline: number analyzed (Participants) | 19
  Bronx baseline | 5.4 (4.4)
  Bronx end: number analyzed (Participants) | 19
  Bronx end | 5.3 (3.8)
  Buffalo baseline: number analyzed (Participants) | 17
  Buffalo baseline | 3.4 (3.7)
  Buffalo end: number analyzed (Participants) | 17
  Buffalo end | 1.3 (2.0)

11. Secondary Outcome: Personal Evaluation of Transitions in Treatment Scale (PETiTP
Description: PETiT is a 30 item self administered scale measuring response to and tolerability and adherence to antipsychotic medication in people with schizophrenia. The range is 30 to 100. Higher scores are better. Although different features are assessed there is a single total score - no subscales.
Time Frame: 8 weeks
Population: 36 subjects entered, 17 at Buffalo and 19 in the Bronx
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 36
score on a scale
  Bronx baseline: number analyzed (Participants) | 19
  Bronx baseline | 43 (9.7)
  Bronx end: number analyzed (Participants) | 19
  Bronx end | 45 (11)
  Buffalo baseline: number analyzed (Participants) | 17
  Buffalo baseline | 46 (11)
  Buffalo end: number analyzed (Participants) | 17
  Buffalo end | 48 (13)

12. Secondary Outcome: Medical Outcomes Study Cognitive Functioning Scale (MOS-COG)
Description: MOS-COG measures day to day problems in six aspects of cognitive functioning. The scores are converted to 0-100 and so can range from 0 to 100 with 100 being the best. Population means are 70 to 80.
Time Frame: 8 weeks
Population: All subjects, 17 at Buffalo, 19 in the Bronx
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 36
score on a scale
  Bronx baseline: number analyzed (Participants) | 19
  Bronx baseline | 17 (5.8)
  Bronx end: number analyzed (Participants) | 19
  Bronx end | 16 (6.3)
  Buffalo baseline: number analyzed (Participants) | 17
  Buffalo baseline | 18 (5.4)
  Buffalo end: number analyzed (Participants) | 17
  Buffalo end | 19 (3.9)

13. Secondary Outcome: Barnes Akathisia Scale
Description: Barnes Akathisia Scale measures akathisia: a score of zero is none (good) maximum score is 12
Time Frame: 8 weeks
Population: All subjects entered, 17 at Buffalo, 19 at Bronx
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 36
score on a scale
  Bronx baseline: number analyzed (Participants) | 19
  Bronx baseline | 0.6 (1.7)
  Bronx end: number analyzed (Participants) | 19
  Bronx end | 0.8 (1.7)
  Buffalo baseline: number analyzed (Participants) | 17
  Buffalo baseline | 1.4 (1.5)
  Buffalo end: number analyzed (Participants) | 17
  Buffalo end | 1.1 (1.7)

14. Secondary Outcome: HbA1c
Description: Lab measure of glycated hemoglobin indicative of blood glucose over the last three months. At that time in the US measured as a percentage (of glucose attached to hemoglobin). No maximum or minimum but over 6.5% is generally considered indicative of diabetes.
Time Frame: 8 weeks
Population: All subjects entered, 19 in the Bronx, 17 at Buffalo
Measure: Mean (Standard Deviation); unit: HbA1c
Arm/Group | Experimental
Number analyzed (Participants) | 36
HbA1c
  Bronx baseline: number analyzed (Participants) | 19
  Bronx baseline | 5.3 (0.6)
  Bronx end: number analyzed (Participants) | 19
  Bronx end | 5.4 (0.7)
  Buffalo baseline: number analyzed (Participants) | 17
  Buffalo baseline | 6.0 (0.9)
  Buffalo end: number analyzed (Participants) | 17
  Buffalo end | 5.7 (0.8)

15. Secondary Outcome: Insulin Level
Description: Measure of the amount of insulin in the blood, in uIU/ml. No minimum or maximum but fasting levels are usually below 25 uIU/ml. After a dose of glucose they may be 30 to 230 uIU/ml.
Time Frame: 8 weeks
Population: All subjects entered, 17 at Buffalo, 19 at Bronx
Measure: Mean (Standard Deviation); unit: uIU/ml
Arm/Group | Experimental
Number analyzed (Participants) | 36
uIU/ml
  Bronx baseline: number analyzed (Participants) | 19
  Bronx baseline | 10 (7.2)
  Bronx end: number analyzed (Participants) | 19
  Bronx end | 13 (14)
  Buffalo baseline: number analyzed (Participants) | 17
  Buffalo baseline | 12 (9.2)
  Buffalo end: number analyzed (Participants) | 17
  Buffalo end | 17 (14)

16. Secondary Outcome: Antipsychotic Medication Costs
Description: No data were collected because it turned out we had no way of measuring the costs.
  No subjects were analysed by costs
Time Frame: 8 weeks
Population: We had no measure of costs, no data were collected
Arm/Group | Experimental
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the time subjects were in the study - screening till 8 weeks on ziprasidone.
Arm/Group | Experimental
Serious Adverse Events (participants affected / at risk) | 1/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=40)
Hospitalization (Psychiatric disorders) | 1 (1) — Relapse of out patient required admission

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No